CLINICAL TRIAL: NCT01193023
Title: Patient-ventilator Asynchrony During Mechanical Invasive Assisted-ventilation in Pediatric Patients
Acronym: NavPed-Inv
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Dr Peter Rimensberger, neonatology and intensive care units, university hospital of Geneva
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HUG-matped 09-253
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Last update posted 2010-09-01 (Estimated); Status verified 2010-08

CONDITIONS: Respiration, Artificial
Keywords: Prospective Studies; Humans, pediatric; Positive-Pressure Respiration/methods*; Respiration, Artificial/methods*; Intensive Care; Intensive Care Units/statistics & numerical data*; Respiration, Artificial/statistics & numerical data*; Patients/statistics & numerical data*; Prevalence; Respiratory Muscles/innervation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pressure support (Active Comparator): in this arm, pressure support will be recorded under 3 conditions:
  * with the initial Expiratory Trigger Setting (ETS)
  * with ETS +10%
  * with ETS -10%
  Interventions: Other: Pressure Support
- NAVA (Experimental): Neurally Adjusted ventilatory Assist is a ventilation mode where the ventilator is piloted by the electrical activity of the diaphragm Ventilation is triggered and cycled off by the electrical activity of the diaphragm, the pressure delivered being proportional to this activity.
  Interventions: Device: NAVA

INTERVENTIONS:
Other: Pressure Support — Ventilation under pressure support
  Arms: Pressure support
Device: NAVA — Ventilation under NAVA
  Arms: NAVA

SUMMARY:
The purpose of this study is to document the prevalence and type of asynchronies incidence during invasive mechanical ventilation in pediatric patients breathing under pressure support.

And to observe the impact of adjusting the expiratory trigger setting on asynchronies, and compare these incidences with asynchronies measured in pediatric patient breathing under NAVA system (Neurally Adjusted Ventilatory Assist).

DETAILED DESCRIPTION:
Two sessions will be recorded, one in PSV, one with NAVA, delivered in a random order after being sure the infant is calm and comfortable, according to his parents and/or the nurse in charge.

Criteria for initiating invasive ventilation and to start PSV will follow the usual practice guidelines of the unit.

Ventilation parameters in PS will be adjusted by the clinician in charge of the patient, as usual based on clinical observation. Investigators will not interfere with ventilator settings. Ventilation will be applied via an endotracheal tube, uncuffed for the majority (if infant < 5 years), according to commonly applied guidelines in this unit.

One 15 minutes session will be recorded, after being sure the infant is calm and comfortable according to the parents and/or the nurse in charge. Then the clinician in charge of the patient will modify the ETS, first decreasing it of 10% below the initial set value, and will be recorded the following 5 minutes after stabilization and secondly increasing it of 10% above the initial set value, and will be recorded the following 5 minutes after stabilization.

NAVA will be set to deliver initially the same peak pressure (comparable level of assist) than during the initial PS period. Same PEEP will be delivered in both modes. This is possible with a pre-visualization window, allowing adjustments before switching to the NAVA mode. Nava ventilation will be recorded during 20 minutes.

The 2 sessions, Pressure support and Nava, will be recorded consecutively.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients from 4 weeks to 12 years (post natal interm infants) admitted to the pediatric intensive care unit (PICU) and receiving mechanical ventilation in pressure support ventilation

Exclusion Criteria:

* Non treated pneumothorax
* Hemodynamic instability
* At least 2 hours following the admission in the PICU in post cardiac surgery
* FiO2 > 0.6
* Poor short term prognosis (defined as a high risk of death in the next seven days)
* contraindication for gastric tube or obtention of a reliable EMGdi signal
* Known esophageal problem (hiatal hernia, esophageal varicosities)
* Active upper gastro-intestinal bleeding or any other contraindication to the insertion of a naso-gastric tube
* Neuromuscular disease
* Patients with a pacemaker

Ages: 4 Weeks to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
asynchronies | 12 months
  Asynchronies during mechanical ventilation are the following: Auto triggering, double triggering, late cycling, premature cycling and ineffective effort.
  all ventilatory parameters are recorded under Pressure support (3 phases: 3 levels of expiratory trigger setting, initial, +10% and -10%, 15 min, 5 min and 5 min respectively) and NAVA (1 phase, 20 min).
  Asynchronies will be determined by measuring each ventilatory cycle of all recordings.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rimensberger, MD, Principal Investigator — Ûniversity hospital of Geneva
Locations (1):
- University hospital of Geneva, Geneva, Switzerland